CLINICAL TRIAL: NCT00983164
Title: Blood Antioxidant Status in Chronic Hepatitis C Patients Before and After Antioxidant Supplementation: a Randomized Clinical Trial
Acronym: HepCAntSup
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Sul de Santa Catarina (Other Government)
Responsible Party: Mirelle Sifroni Farias, Universidade Federal Santa Catarina
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 120/07 CEP; 120/07 CEP
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Hepatitis C; Oxidative Stress
Keywords: antiviral therapy; antioxidant therapy; hepatitis C virus; oxidative stress; vitamin E
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- group I (No Intervention): group I - controls
- group II (Experimental): group II - patients with hepatitis C without treatment
  Interventions: Dietary Supplement: Antioxidant Supplementation
- group III (Experimental): group III - patients with hepatitis C treated weekly with pegylated interferon combined with daily ribavirin
  Interventions: Dietary Supplement: Antioxidant Supplementation

INTERVENTIONS:
Dietary Supplement: Antioxidant Supplementation — antioxidant supplementation (vitamin E 800 mg, C 500 mg and zinc 40 mg) for 24 weeks
  Arms: group II; group III

SUMMARY:
The objective of the present study is to evaluate the antioxidant status in the blood of HCV patients treated with pegylated interferon (2a 1.5 ug/kg; 2b 180 ug) combined with ribavirin (1000 to 1250 mg) before and after supplementation of vitamins E, C and the mineral zinc (800 mg,500 mg and 40 mg; respectively) during six months.

DETAILED DESCRIPTION:
The WHO estimated that around 170 million people are infected by HCV, about 3% of the world population. HCV is the leading cause of acute hepatitis and chronic liver disease, which may lead to cirrhosis and hepatocellular carcinoma.

The combined therapy with interferon with or without pegylation associated with ribavirin has shown greater sustained virological response than monotherapy with interferon-alpha, however this response still represents around 60% of cases. The mechanisms by which HCV causes cellular damage are not yet well understood, however immune liver damage, direct cytotoxic damage mediated by different viral products and also oxidative stress have been implicated in the pathogenesis of chronic hepatitis C. Several studies support that reactive oxygen species (ROS) and oxidative stress are involved in the pathogenesis of hepatitis C, despite that increased ROS levels in HCV patients might be beneficial by suppressing HCV replication. ROS are involved in several diseases and cause oxidative damage to lipids, DNA, proteins and carbohydrates.

ELIGIBILITY:
Inclusion Criteria:

* without the presence of illnesses associated with systemic diseases, no chronic alcoholism, without HIV coinfection, and were not participating in other studies.
* Patients with hepatitis C were selected according to the Clinical Protocol and Guidelines for Therapeutic Hepatitis C Viral.
* Group I - All subjects were negative for HCV, HBV, HIV, HBsAg, anti-HBc total, anti-HCV and normal serum transaminases.

Exclusion Criteria:

* Patients with one of the following laboratory abnormalities were also excluded: leukocytes, neutrophils, platelets, serum creatinine 1.5 times upper limit of normal, elevated thyroid stimulating hormone, alpha-fetoprotein above normal limits, and/or focal lesion on ultrasound performed within 1 month of study entry.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mirelle Sifroni Farias, Principal Investigator — Universidade Federal Santa Catarina
Locations (3):
- Brazil (3):
  - Hospital Nereu Ramos, Florianópolis, Santa Catarina
  - Hospital Universitário Universidade Federal Santa Catarina, Florianópolis, Santa Catarina
  - Policlínica II, Florianópolis, Santa Catarina